CLINICAL TRIAL: NCT04995237
Title: Richmond Health and Wellness Program (RHWP) Prescription Produce Plan (PPP) Pilot Study
Brief Title: RHWP Prescription Produce Plan
Acronym: PPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20022162
Record Dates: First submitted 2021-07-30; First posted 2021-08-06 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Quality of Life

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prescription Produce Plan (PPP) (Experimental): PPP provides access to fresh produce along with individual goal setting and education
  Interventions: Behavioral: PPP

INTERVENTIONS:
Behavioral: PPP — Participants will be provided with a weekly bag of produce, information about how to cook the produce, assistance in setting quality of life goals, and individualized teaching to support meeting participant's set goals.

SUMMARY:
The purpose of this research study is to find out if access to fresh produce along with individual goal setting and education influences vegetable consumption, self-management [self-efficacy], resilience, or quality of life. Researcher think access to fresh produce along with individual goal setting and education, may improve all of the above. This study will allow them to learn more about it.

DETAILED DESCRIPTION:
This research study focused on examining how a Prescription Produce Plan (PPP) may influence vegetable consumption, self-management [self-efficacy], resilience, and quality of life in older adults. This research study involves meeting with a team of VCU students and faculty to learn information about nutrition.

In this study, participants will be asked to do the following things:

1. Complete a total of five (5) surveys and the consent process during the enrollment visit lasting approximately 30 to 60 minutes.
2. Record their blood pressure readings and blood glucose readings [if they already do this] once a week in a notebook provided by the research team and then self-report the blood pressure and blood glucose readings at the next two (2) study visits.
3. Receive individualized teaching supporting obtaining the goals at this visit and future study visits. The study team will discuss with participants the contents of the produce bags and how to cook the contents of the bag. They will also work with participants to set goals for themselves. Goals for this study will focus on vegetable consumption, weight management, and either blood pressure and/or blood glucose measurements. The initial study visit may last approximately 30 minutes.
4. At the end of the initial study visit, you will receive a voucher from the Shalom Farms Mobile Market for once a week redemption over the course of 6 weeks while participating in the program. VCU Health Hub 25th Street participants will receive a produce bag at the end of this visit and will need to come to the Health Hub weekly to pick up the produce bag.
5. Subsequent study visits will focus on participant goals. Participants will meet with the study team to discuss if goals were met or not met and the study team will provide individualized teaching to support meeting participant's set goals. The study team will ask participants to meet with them twice after the initial study visit for approximately 20 to 30 minutes at each visit. These meetings will be at Week #3 and at Week #6.
6. Participants will record in provided notebooks their blood pressure, weight, and blood glucose [if they are already checking their blood glucose prior to participating in this study]. These measurements will also be reported during study visits.
7. Participants are asked to meet with a member of the research team after six (6) weeks of participating in the study to complete a total of three (3) post-study surveys. This visit will last approximately 30 minutes.

Participation in this study will last up to 8 weeks for a total of approximately 3 hours of in person visits. Approximately 30 individuals will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Richmond Health Wellness Program [RHWP]Participant or interested in joining RHWP
* age 40 and older
* live in Richmond
* have a desire to set goals having access to fresh produce

Exclusion Criteria:

• not interested in joining Richmond Health and Wellness Program

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Change in number of vegetable servings consumed | Baseline to 6 weeks
  At each study visit, participants will self report average number of vegetable servings consumed daily.
Number of participants who met weight management goals | 6 weeks
  At each study visit, participants will self report whether or not they met their weight management goal which they set during the previous study visits.
Number of participants who met blood glucose levels goals | 6 weeks
  For participants who already monitor their blood glucose, at each study visit, participants will self report whether or not they met their glucose level goals which they set during the previous study visits
Number of participants who met blood pressure reduction goals | 6 weeks
  At each study visit, participants will self report whether or not they met their blood pressure reduction goal which they set during the previous study visits.
Number of participants who feel healthier | 6 weeks
  At each study visit, participants will be asked if they feel healthier (yes or no).

SECONDARY OUTCOMES:
Change in self-reported blood pressure reading | Baseline to 6 weeks
  Participants will be provided with an automatic blood pressure machine, shown how to use it with, and given a handout with instructions on how to record and monitor their blood pressure at home. Participant will self-report the results of their blood pressure reading during the study visits.
Change in self-reported blood glucose reading | Baseline to 6 weeks
  For participants who already monitor their blood glucose, participants will self-report the results of their blood glucose reading during the study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Battle, PhD, RN, FNP-BC, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT04995237/ICF_000.pdf